CLINICAL TRIAL: NCT06982001
Title: Importance of Arterial Measurement Sites on Intraoperative Hemodynamic Management of Major Abdominal Surgeries and Artificial Intelligence-based Prediction of Arterial Gradient Using Peripheral Radial Pressure Waveform Analysis
Brief Title: ImPortance of Arterial Measurement Sites (IPAMS) on Intraoperative Hemodynamic Management
Acronym: IPAMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Fondation Anesthesiologistes du Quebec (Unknown); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-3299
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-10

CONDITIONS: Perioperative Care; Hemodynamics; Monitoring Blood Pressure; Arterial Lines; Anesthesia; Vasopressor; Fluid Management; Artificial Intelligence in Operating Room; Artificial Intelligence (AI)
Keywords: Comparison of arterial catheterization sites on hemodynamic monitoring; Incidence of radial-brachial pressure gradient; Risk factors of radial-brachial pressure gradient; Effect of arterial catheterization sites on hemodynamic management; Effect of peripheral vs central arterial pressure measurements in intraoperative hemodynamic management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brachial artery-guided interventions (Experimental): In this experimental group, hemodynamic management will be guided by using the brachial arterial line. Both a radial and a brachial line will be inserted for simultaneous monitoring, but the anesthesiologist will only see the brachial arterial line and will guide his drug administration and hemodynamic management on the brachial measurements.
  Interventions: Behavioral: Brachial line guided hemodynamic management; Device: Radial line catheterization; Device: Brachial line catheterization
- Radial artery-guided interventions (Active Comparator): In this group, hemodynamic management will be guided by using the radial arterial line. Both a radial and a brachial line will be inserted for simultaneous monitoring, but the anesthesiologist will only see the radial arterial line and will guide his drug administration and hemodynamic management on the brachial measurements.
  Interventions: Behavioral: Radial line guided hemodynamic management; Device: Radial line catheterization; Device: Brachial line catheterization

INTERVENTIONS:
Behavioral: Brachial line guided hemodynamic management — Anesthesiologists in charge of the patients will guide their hemodynamic management based on the monitoring of brachial/humeral arterial line, instead of the most frequently used radial line.
  Arms: Brachial artery-guided interventions
Behavioral: Radial line guided hemodynamic management — The anesthesiologist will guide their hemodynamic management on the classically used radial arterial line.
  Arms: Radial artery-guided interventions
Device: Radial line catheterization — An arterial line will be inserted in the radial artery of the patient.
Device: Brachial line catheterization — An arterial line will be inserted in the brachial artery of the patient.

SUMMARY:
The goal of this clinical trial is to demonstrate the importance of arterial pressure measurement sites during major abdominal surgeries. This randomized controlled trial will compare arterial pressure measurements obtained from radial artery catheterization (the current standard method of monitoring) with those obtained from brachial artery catheterization (a more accurate reflection of central arterial pressure). At the end of the study, we are looking to answer the following questions:

1. Does arterial pressure measurement sites influence the amount of vasopressors that is administered during major abdominal surgeries?
2. What are the instances where there is a difference between peripheral (radial catheter) and central (brachial catheter) monitoring and what are the risk factors leading to the appearance of this radial-brachial pressure gradient?
3. With the data collected, can artificial intelligence based analysis help predict the reliability of a radial monitoring and help guide clinicians on choosing a peripheral versus central arterial pressure monitoring site? All adult participants who are scheduled for elective major abdominal surgeries and meeting our inclusion criteria will be approached and included if they consent. Participants will be randomized 1:1 in the intervention group and the standard of care group. In the intervention group, the brachial arterial line will be used intraoperatively to guide vasopressor and fluid administration. A radial line will also be installed to measure the radial arterial pressure simultaneously, but will not be used to guide hemodynamic management. In the standard of care group, both lines will be installed just like in the intervention group, however, it is the radial arterial line that will guide fluid and vasopressor administration. In both groups, the anesthesia protocol will be standardized and the anesthesiologist will be blinded to the arterial pressure measurement site.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 90 years of age;
* Major abdominal surgery via laparoscopy or laparotomy under general anesthesia - with or without concomitant use of regional or neuraxial anesthesia;
* Expected anesthesia time of more than 120 minutes.

Exclusion Criteria:

* Known peripheral severe vascular disease with subclavian artery stenosis,
* Significant arterial gradient between arms with preoperative non-invasive bloop pressure measurements (>25 mm Hg of systolic blood pressure or 10 mm Hg of mean arterial pressure);
* Inability or contraindications to insert arterial line on either arm (arteriovenous fistula, surgical sterility);
* Known allergies, intolerance, other medical conditions that precludes the use of prescribed general anesthesia protocol for this trial;
* Inability to communicate in French or English.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average administration of noradrenaline | Intraoperative administration
  The administration of norepinephrine will be continuously monitored during the surgery, and the time-weighted dose per kilograms will be extracted between the surgical incision and the last skin suture.

SECONDARY OUTCOMES:
Total amount of noradrenaline administered | Intraoperative administration
  Total dose of norephinephrine from skin incision to skin suture.
Total time of hypotension | Intraoperative
  Total time and time weighted spent below the inferior threshold (baseline MAP-20%), measured independently by the radial line and the brachial line.
Occurrence and depth of radial-to-brachial gradient | Intraoperative
  The depth-weighted time spent with a pressure gradient between the radial and brachial arterial pressures
Dose of other inotropes and vasopressors | Intraoperative administration
  Any administration of vasopressor or inotropes, other than the noradrenaline measured in the primary outcome. Total dose and time weighted if perfused.
Fluid balance | Intraoperative administration
  Total and time weighted fluid administered intraoperatively (volume and nature)
Urine output | Intraoperative
  Total and time weighted output of urine, measured every hour
Total consumption of opioids | Intraoperative
  Total and time weighted dose of opioids (remifentanil) administered intraoperatively
Total consumption of hypnotic drug | Intraoperative
  Total and time-weighted dose of hypnotic drug administered.
Cumulative duration of burst suppression and low BIS values | Intraoperative
  Total, time weighted and importance weighted duration of BIS value below 40, and total and time-weighted duration of burst suppression (suppression time).
Troponin and Creatinine lab measurements | Post-anesthesia care unit and post-operative day 1,3 and 7
  Value of troponin and creatinine of the patient
Clavien-Dindo Score | Post-operative day 1,3 and 7
  A validated score evaluating the occurence of post-operative complications.
Composite occurence of postoperative complications | Post-operative day 1,3 and 7
  Composite outcome comprising the occurrence of myocardial injury after non-cardiac surgery (MINS), stroke, arrythmia, and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
IPD might not be shared depending on the ethical consideration of sharing the information. We are currently working on a central database for perioperative research data collected at our institution, which will structure all IPD. Depending on the advancement of this initiative, we might enable IPD.

REFERENCES:
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Galluccio ST, Chapman MJ, Finnis ME. Femoral-radial arterial pressure gradients in critically ill patients. Crit Care Resusc. 2009 Mar;11(1):34-8. PMID 19281442
- [Background] Ahuja S, Mascha EJ, Yang D, Maheshwari K, Cohen B, Khanna AK, Ruetzler K, Turan A, Sessler DI. Associations of Intraoperative Radial Arterial Systolic, Diastolic, Mean, and Pulse Pressures with Myocardial and Acute Kidney Injury after Noncardiac Surgery: A Retrospective Cohort Analysis. Anesthesiology. 2020 Feb;132(2):291-306. doi: 10.1097/ALN.0000000000003048. PMID 31939844
- [Background] Renaud-Roy E, Stockle PA, Maximos S, Brulotte V, Sideris L, Dube P, Drolet P, Tanoubi I, Issa R, Verdonck O, Fortier LP, Richebe P. Correlation between incremental remifentanil doses and the Nociception Level (NOL) index response after intraoperative noxious stimuli. Can J Anaesth. 2019 Sep;66(9):1049-1061. doi: 10.1007/s12630-019-01372-1. Epub 2019 Apr 17. PMID 30997633
- [Background] Tang Y, Zhu C, Liu J, Wang A, Duan K, Li B, Yuan H, Zhang H, Yao M, Ouyang W. Association of Intraoperative Hypotension with Acute Kidney Injury after Noncardiac Surgery in Patients Younger than 60 Years Old. Kidney Blood Press Res. 2019;44(2):211-221. doi: 10.1159/000498990. Epub 2019 Mar 29. PMID 30928979